CLINICAL TRIAL: NCT00614302
Title: Italian Prospective Data Collection for Better Patient Characterization in a Highly Treatment Experienced Patient Population
Brief Title: Italian Prospective Data Collection for Better Patient Characterization in a Highly Treatment Experienced Population
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 1182.130
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: TPV

SUMMARY:
Data collection for better patient characterization in a highly treatment experienced population. Studying the clinical practice for the treatment of HIV multiexperienced patients in the real life.

The research will be divided into two phases:

* The first phase intends to define and understand the clinical practice using a questionnaire about general topics: definitions of multiexperienced patients and VL failure, therapeutic strategies and behaviour in particular cases.
* The second part of the research will collect the clinical data of double PIs failure patients.

ELIGIBILITY:
Inclusion Criteria:

Patients double PIs failure

Exclusion Criteria:

Not Applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients
Sampling Method: Non-Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To study in the clinical practice the choice of a specific salvage regimen for multiexperienced patients. | 48 weeks

SECONDARY OUTCOMES:
Reason of each VL failure or switching | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (21):
- Italy (21):
  - Boehringer Ingelheim Investigational Site, Ancona
  - Boehringer Ingelheim Investigational Site, Bari
  - Boehringer Ingelheim Investigational Site, Benevento
  - Boehringer Ingelheim Investigational Site, Bisceglie
  - Boehringer Ingelheim Investigational Site, Bologna
  - Boehringer Ingelheim Investigational Site, Brescia
  - Boehringer Ingelheim Investigational Site, Busto
  - Boehringer Ingelheim Investigational Site, Caserta
  - Boehringer Ingelheim Investigational Site, Catania
  - Boehringer Ingelheim Investigational Site, Cremona
  - Boehringer Ingelheim Investigational Site, Florence
  - Boehringer Ingelheim Investigational Site, Genova
  - Boehringer Ingelheim Investigational Site, Legnano
  - Boehringer Ingelheim Investigational Site, Milan
  - Boehringer Ingelheim Investigational Site, Napoli
  - Boehringer Ingelheim Investigational Site, Padua
  - Boehringer Ingelheim Investigational Site, Palermo
  - Boehringer Ingelheim Investigational Site, Pavia
  - Boehringer Ingelheim Investigational Site, Roma
  - Boehringer Ingelheim Investigational Site, Sassari
  - Boehringer Ingelheim Investigational Site, Torino